CLINICAL TRIAL: NCT02398864
Title: Accuracy and Safety of Endobronchial Ultrasound (EBUS) in Suspected Non-malignant Mediastinal Lymphadenopathy
Acronym: EBUS-nonM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1203-2015
Record Dates: First submitted 2015-03-13; First posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Mediastinal Lymphadenopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- endobronchial ultrasound bronchoscopy (Experimental): EBUS with TBNA
  Interventions: Procedure: EBUS with TBNA

INTERVENTIONS:
Procedure: EBUS with TBNA — endobronchial ultrasound (EBUS) with transbronchial needle aspiration (TBNA)

SUMMARY:
To examine whether EBUS with transbronchial needle aspiration (TBNA) can accurately and safely diagnose enlarged lymph nodes in the chest in patients without suspected malignancy

DETAILED DESCRIPTION:
There is no single method to investigate mediastinal LN invasion. Hence, a patient may have to undergo several tests and procedures. Noninvasive and invasive approaches are employed. Within the invasive techniques, endoscopic ultrasonography with needle aspiration (EUS-FNA) and endobronchial ultrasonography with transbronchial needle aspiration (EBUS-TBNA) are gaining importance in mediastinal staging. Endobronchial Ultrasound (EBUS) is a procedure that is performed via flexible bronchoscopy under moderate sedation for visualization of lymph nodes in the chest and biopsy under real-time guidance usually for the staging of lung cancer or evaluation of enlarged lymph nodes. In addition, lung lesions or masses can be visualized and biopsied in the same sitting. The use of EBUS has enhanced the safety and diagnostic yield of flexible bronchoscopy. It provides ultrasonographic images and permits needle aspiration under direct vision for cytology specimen analysis. As more evidence is being accumulated on these staging approaches, the number of cervical mediastinoscopies, considered as the gold-standard for mediastinal staging, is diminishing.

ELIGIBILITY:
Inclusion Criteria:

* adults (18 Years and older) with mediastinal lymphadenopathy.

Exclusion Criteria:

* known or suspected malignancy
* no informed consent
* pts with anterior mediastinal lesions
* contraindications to EBUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of EBUS-diagnosis | 2 years
  Sensitivity defined as the proportion of participants with a positive EBUS-diagnosis accordant to final diagnosis, specificity, positive predictive value, negative predictive value and accuracy will be determined

SECONDARY OUTCOMES:
Risk factors related with the development of complications | 2 years
  1. Complications during procedure as Bleeding, pneumothorax, shock cardiac arrhythmia, change of oxygen desaturation
  2. Complication after procedure as fever, mediastinitis, bleeding, pneumothorax and other complications after 24hr
Risk factors related with the procedure | 2 years
  1. dosage of sedative drugs
  2. Procedure time
  3. Total aspiration number
  4. Location of sampled lymph node
  5. Sampling number of lymph nodes
  6. the development of comorbidities
  7. Pulmonary function tests

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Fuehner, MD, Principal Investigator — Hannover Medical School